CLINICAL TRIAL: NCT06908278
Title: The Impact of Simulation-Based Education on Midwifery Students' Episiotomy Self-Efficacy Levels: A Randomized Controlled Trial
Brief Title: The Impact of Simulation-Based Education on Midwifery Students' Episiotomy Self-Efficacy Levels
Acronym: SBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Zeynep Ogul, Assit. Prof, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 51.2024fbu
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Episiotomy; Self Efficacy; Simulation Based Medical Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm 1: Suture Simulation Training (Experimental): Participants in this arm will receive suture simulation training for episiotomy repair. This includes both theoretical instruction and hands-on practice using a suture simulator in a controlled, guided setting. The purpose of this intervention is to enhance self-efficacy and competence in episiotomy suturing.
  Interventions: Behavioral: Suture Simulation Training for Episiotomy Repair
- Experimental Arm 2: Sponge Simulation Training (Experimental): Participants in this arm will receive sponge simulation training for episiotomy repair. The training includes theoretical education followed by hands-on practice using sponge materials that mimic soft tissue. The goal is to develop suturing skills and improve participants' self-efficacy in performing episiotomy repairs in a safe and controlled environment.
  Interventions: Behavioral: Suture Simulation Training for Episiotomy Repair

INTERVENTIONS:
Behavioral: Suture Simulation Training for Episiotomy Repair — This intervention involves training participants to perform episiotomy repairs using a suture simulator. Participants will practice suturing techniques in a controlled, safe environment to improve their self-efficacy in performing the procedure. The training includes both theoretical learning and hands-on practice. The goal is to enhance the participants' confidence and competence in performing episiotomies.
  (This description outlines the nature of the intervention and the learning objectives.)

SUMMARY:
Problem: Self-efficacy, the belief in one's ability to perform tasks, plays a critical role in learning. Inadequate self-efficacy can hinder the development of essential clinical skills in midwifery students.

Background: Simulation-based education provides a safe learning environment that enhances students' skills and confidence without the fear of mistakes. However, the comparative effectiveness of different simulation methods on self-efficacy remains unclear.

Aim: This randomized controlled trial aims to evaluate the effectiveness of suture simulation training versus sponge simulation training on midwifery students' self-efficacy in episiotomy repair. Specifically, it seeks to answer the following questions:

Does suture simulation training improve self-efficacy in episiotomy repair more effectively than sponge simulation training?

What challenges or difficulties do students encounter with each simulation method?

Methods: A total of 84 midwifery students participated in the study. They were randomly assigned to two groups:

Intervention 1 (n=42): Practiced on a suture simulator.

Intervention 2 (n=42): Practiced on a sponge simulator.

Both groups received identical theoretical training on episiotomy repair through slide presentations and video demonstrations over two sessions lasting four hours. Students:

Engaged in hands-on training with their assigned simulation method for four weeks.

Attended clinic visits every two weeks for skill assessments and feedback.

Maintained a self-report diary documenting their confidence levels and skill progression.

Data collection included demographic characteristics, self-efficacy assessments using the Episiotomy Skills Self-Efficacy Scale (ESSES), and observational data. Statistical analyses were planned using t-tests and chi-square tests, with significance set at p<0.05.

Future results will be analyzed and reported separately in the Results Section, following data collection and processing.

ELIGIBILITY:
Inclusion Criteria:

Ability to communicate in Turkish.

Enrollment in the midwifery department.

Registration in courses on midwifery care for high-risk pregnancies and postpartum care following high-risk deliveries.

Exclusion Criteria:

Inability to communicate in Turkish.

Not enrolled in the midwifery department.

Not registered in the relevant courses.

Any condition preventing participation in hands-on simulation training.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
Change in Self-Efficacy Scores for Episiotomy Repair | Baseline (pre-training), immediately after training, and 4 weeks post-training
  Self-efficacy in episiotomy repair will be assessed using the Episiotomy Skills Self-Efficacy Scale (ESSES). The ESSES is a validated instrument measuring students' confidence in performing episiotomy repair. Scores range from 0 to 100, with higher scores indicating greater self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahce University, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No